CLINICAL TRIAL: NCT03427437
Title: Ultrasound-Guided Versus Conventional Method for Caudal Block in Children
Brief Title: Ultrasound-Guided Versus Conventional Method for Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Karaca (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, Omer Karaca, Medical Doctor, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 16/354
Record Dates: First submitted 2018-01-23; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Ultrasound Therapy; Complications
Keywords: sacral canal; sacral hiatus; ultrasound
MeSH Terms: interventions — Bupivacaine; Epinephrine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Group (Active Comparator): Caudal block was performed by conventional method with %0,25 bupivacaine plus 1/200.000 adrenalin
  Interventions: Drug: Bupivacaine; Drug: Adrenalin
- Ultrasound Group (Active Comparator): Caudal block was performed by ultrasound method with %0,25 bupivacaine plus 1/200.000 adrenalin
  Interventions: Drug: Bupivacaine; Drug: Adrenalin; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine — caudal block was performed by conventional and ultrasound method with %0,25 bupivacaine + 1/200000 adrenalin
  Other Names: Bustesin,Vem Drug, Ankara, Turkey
Drug: Adrenalin — caudal block was performed by conventional and ultrasound method with %0,25 bupivacaine + 1/200000 adrenalin
  Other Names: Adrenalin 0.5 mg, Osel Drug, Istanbul, Turkey
Device: Ultrasound — caudal block was performed by ultrasound method
  Other Names: Sonosite M Turbo, USA
  Arms: Ultrasound Group

SUMMARY:
Caudal epidural block has been widely used, especially in pediatric surgery, to supply intraoperative and postoperative analgesia by affecting the region between T10 and S5 dermatomes in surgeries below the umbilical level.

In conventional single-shot caudal block, the needle is inserted through the skin with a 60-80 degrees angle, until the sacrococcygeal ligament is passed through. Then the angle of the needle is decreased to 20-30 degrees and inserted further for an additional 2-3 mm, entering into the sacral canal.There is a risk of dural or vascular puncture when the needle is passing through sacral canal. Other complications are the soft tissue bulging, intraosseous injections and systemic toxicity.

Many anatomical variations have been reported for sacral hiatus and sacral cornua. Therefore, the success rate of the classic caudal epidural anesthesia method in pediatric patients has been reported to be about 75%.

With the usage of ultrasonography in regional anesthesia, many advantages have been reported. In particular ultrasonography under longitudinal image is helpful for visualization of the sacral hiatus, sacrococcygeal ligament, duramater, epidural space and the distribution of the local anesthetic agent Therefore, this significantly increases the block success and visualization of where local anesthetic is injected.

The primary aim of this study was compare the success rate of ultrasound guided sacral hiatus injection and conventional sacral canal injection. Secondary objectives are; block performing time, number of needle puncture, success at first puncture and complication rate. However age and weight encountered wtih these complications are registered.

DETAILED DESCRIPTION:
The caudal block was performed in Group C by via conventional methods. The sacral cornus and the sacral hiatus were palpated. After sterilization of the region, a 22- gauge caudal needle was inserted into the skin with at a 60-80 degree angle and until the sacrococcygeal ligament was passed punctured, as determined with by a "popping sensation." feeling (puncture of the sacrococcygeal ligament). Then, the angle of the needle was then reduced to 20-30 degrees and inserted further for an additional 2-3mm, entering into the sacral canal. After verifingverifying the absence of any blood or cerebrospinal fluid in the aspiration, a test dose of 0.1 ml/kg of local anesthetic (LA) with adrenalin at a ratio of 1: 200000 was injected under hemodynamic and ECG monitoring. Following a negative test dose, the rest of the LA was slowly injected slowly over 1 min. In the case of the needle touching the bony tissue, blood aspiration, or bulging into of the subcutaneous tissue, the angle of the needle was changed and the intervention was repeated.

The caudal block was performed by via ultrasound guided ultrasound guidance in Group U. After sterilization of the region and using ultrasound guidanceUSG with a sterile plastic cover and gel, the sacral hiatus was visualized via an out-of-plane technique at the level of the sacral cornus at the out of plane via the lineerlinear transducer of an M-Turbo ultrasound machine (TM; Fujifilm SonoSite Inc., (Washington, WA, United StatesUSA) ultrasound machine at 13 MHz, and the, depth and gain was adjusted to for optimal visual quality. The ultrasound ultrasound transducer was first placed transversely at the midlain midline to obtain the transvers view of the two cornua, the sacrococcygeal ligament, the sacral bone, and the sacral hiatus. At this level, the ultrasound ultrasound transducer was rotated 90 degrees to obtain the longitudinal view of the sacrococcygeal ligamantligament and sacral hiatus, and was then placed between the two cornua. A 22- gauge caudal needle was advanced toward the upper third of the sacrococcygeal ligament. The needle advancement was terminated right after penetrating the sacrococcygeal ligament. At this level, after confirming the absence of any blood or cerebrospinal fluid in the aspiration and a negative test dose, the rest of the LA was injected over 1 min under while observing the ultrasound ultrasound longitudinal image

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologist) I children aged between 6 months and 8 years old who underwent elective hypospadias, circumcision and both surgery

Exclusion Criteria:

* Severe systemic disease, previous neurological or spinal disorder, coagulation anomaly, allergy against local anesthetics, local infection at block site or with a history of premature birth

Ages: 6 Months to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
success rate of block | Intraoperative period
  absence of significant motor movements following surgical induction or aberrations in heart and or respiratory rates

SECONDARY OUTCOMES:
block performing time | Intraoperative first hour
  The block time was defined as the period between the insertion of the needle and termination of local anesthetic administration
first puncture success rate | Intraoperative first hour
  The first puncture success rate was defined as reaching the sacral canal or sacral hiatus with a single-needle orientation on the first puncture without any withdrawal from the skin.
complications | Intraoperative first hour
  situations such as vascular puncture, bone contact, subcutaneous injection encountered, when the caudal block was performed,
age and weight encountered complications | Intraoperative first hour
  below which age and weight

CONTACTS AND LOCATIONS:
Overall Officials: Omer Karaca, MD, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang LZ, Hu XX, Zhang YF, Chang XY. A randomized comparison of caudal block by sacral hiatus injection under ultrasound guidance with traditional sacral canal injection in children. Paediatr Anaesth. 2013 May;23(5):395-400. doi: 10.1111/pan.12104. Epub 2012 Dec 29. PMID 23278906
- [Result] Ahiskalioglu A, Yayik AM, Ahiskalioglu EO, Ekinci M, Golboyu BE, Celik EC, Alici HA, Oral A, Demirdogen SO. Ultrasound-guided versus conventional injection for caudal block in children: A prospective randomized clinical study. J Clin Anesth. 2018 Feb;44:91-96. doi: 10.1016/j.jclinane.2017.11.011. Epub 2017 Nov 21. PMID 29161549